CLINICAL TRIAL: NCT06544174
Title: Long-term Clinical Follow-up After PCI for CTO
Acronym: LT-CTO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01-008 LECLERCQ
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Coronary Total Occlusion
Keywords: CTO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successful CTO-PCI: Success was defined as a procedure achieving a final residual stenosis < 30% (by visual estimation) and a TIMI flow grade 3 after CTO recanalization in all living patients within 24h following angioplasty.
  Interventions: Other: Percutaneous Coronary Intervention of CTO
- Failed CTO-PCI: Success was defined as a procedure achieving a final residual stenosis < 30% (by visual estimation) and a TIMI flow grade 3 after CTO recanalization in all living patients within 24h following angioplasty.

INTERVENTIONS:
Other: Percutaneous Coronary Intervention of CTO — CTO-PCI is a procedure of interventional cardiology attempting revascularisation of the CTO
  Groups: Successful CTO-PCI

SUMMARY:
The research aimed to evaluate the impact of a successful Percutaneous coronary intervention of chronic total occlusions (CTO-PCI) on long-term MACE (Major Cardiovascular Events), symptoms, survival, Left Ventricular Ejection Fraction (LVEF) and myocardial ischemia up-to-8-years follow-up.

DETAILED DESCRIPTION:
With this observational and prospective study, this research aimed to evaluate the impact of a successful CTO-PCI on long-term MACE (Major Cardiovascular Events), symptoms, survival, LVEF and myocardial ischemia up-to-8-years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* who underwent at least one CTO procedure between 2025 and 2022 in Montpellier University Hospital
* symptomatic of reversible myocardial ischemia
* proof of myocardial viability

Exclusion Criteria:

* refusal of the patient to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent an attempt of percutaneous recanalization of a CTO at Montpellier University Hospital between January 2015 and December 2022. All patients had symptoms (angina or dyspnea) and/or reversible myocardial ischemia in the territory of the occluded artery and myocardial viability
Sampling Method: Non-Probability Sample
Enrollment: 448 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Major cardiovascular events (MACE) | Up to 8 years
  Incidence of composite of cardiac death, non-fatal myocardial infarction and new target vessel revascularization

SECONDARY OUTCOMES:
Non combined MACE components | Up to 8 years
  Incidence of Cardiac death, non-fatal myocardial infarction and new target vessel revascularization
In-hospital events | Up to one week
  Incidence of Procedural complications including death, periprocedural MI, coronary perforation, pericardial tamponade requiring drainage, local vascular complications, major bleeding, contrast induced nephropathy, stroke
Restenosis | Up to 8 years
  Incidence of Restenosis Defined as a greater than 50% diameter stenosis at follow-up angiogram of the first dilated total occlusion. Reocclusion was defined as recurrent total occlusion of the first dilated total occlusion.
Ischemic burden | Up to 8 years
  Comparison between pre and post-CTO ischemic tests
Stent thrombosis | Within 30 days after the procedure
  Incidence of stent thrombosis defined as any myocardial infarction with angiographic confirmation of in-stent thrombus or unexplained death
LVEF | Up to 8 years
  Percentage of Increase or decrease in LVEF after the CTO procedure compared with baseline LVEF

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, PU-PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No